CLINICAL TRIAL: NCT01816451
Title: Physiological Responses to Constant-load (Continuous) vs. Variable-intensity (Interval) During 14 Weeks of Supervised Aerobic Exercise on Active Men.
Brief Title: Physiologic Adaptations to Interval and Continuous Running at Low Volume and Vigorous Intensity Over 14-Weeks.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trás-os-Montes and Alto Douro (Other)
Responsible Party: Principal Investigator, Laura Castro de Garay, Principal Investigator, University of Trás-os-Montes and Alto Douro
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: UFRJ-2010
Record Dates: First submitted 2013-03-14; First posted 2013-03-22 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Exhaustion - Physiological
Keywords: aerobic capacity; cardiorespiratory training; blood lactate concentration; heart rate
MeSH Terms: interventions — Stochastic Processes; Jogging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- interval (Experimental): The running training for interval group were performed on a treadmill for a period of 14 weeks, with a frequency of three times a week, lasting 20-minutes per session thus completing 46 sessions of training. The intensity and volume of training both were adapted according to the recommendations of the American College of Sports Medicine. The interval training group intensities ranged between 84-87% of maximal heart rate (HRmax) (vigorous intensity), 88-93%HRmax (near maximum intensity) and 94-99% HRmax (maximum intensity).
  Interventions: Other: running training
- continuous (Experimental): The running training for continuous group were performed on a treadmill for a period of 14 weeks, with a frequency of three times a week, lasting 20-minutes per session thus completing 46 sessions of training. The intensity and volume of training both were adapted according to the recommendations of the American College of Sports Medicine.The continuous group ran at an intensity of ~87% of maximal heart rate (HRmax)
  Interventions: Other: running training
- control (No Intervention): The control group did not do the running training program. Control did their normal physical activities.

INTERVENTIONS:
Other: running training — The present study was designed to compare the physiological effects between the two training regimes and the control group.The subjects from interval and continuous group performed others activities as resistance training, swimming or soccer. Those activities wasn't controlled by our study, but the individual didn't do physical activities at least 3 hours before started our running sessions. The control group simply performed their normal physical activities (resistance training, swimming or soccer). But, each 3 weeks we had a contact with control group to check about any injury or illness that could affect the final results. None were found.
  Other Names: Stochastic; aerobic; run
  Arms: continuous; interval

SUMMARY:
The purpose of this study was to verify physiological responses to constant-load (continuous) vs. variable-intensity (interval) during 14 weeks of aerobic exercise on active men. The hypothesis was that would be differences in physiological variables on distinct modes of execution performed on the treadmill over a period of 14 weeks of training.

DETAILED DESCRIPTION:
Initially there were thirty five subjects, but due factors outside the present study, three individuals were excluded from the program. Two individuals during maximal exercise test (VO2) showed clinical impairment test being interrupted by the doctor and the third individual presented a plantar fasciitis in the early familiarization. Thirty two healthy and active males volunteered to participate in the study. All subjects exercised habitually, with at least 1 year experience aerobic training. The Human Ethics Committee of Rio de Janeiro Federal University approved this study (no 58659/02471312.8.0000.5257).The subjects performed a total of nine visits to the laboratory of the Brazilian Navy at City of Rio de Janeiro for physical tests on different days, except between visits I-II and VII-III. The interval between visits was one week between visits II-III-IV and VIII-IX, six weeks between the first day of training and visits V, four weeks between V-VI-VIII. All subjects from interval and continuous groups performed a total of 46 sessions of supervised running program.

ELIGIBILITY:
Inclusion Criteria:

* self reporting no contraindication to high-intensity exercise.
* physically active on cardiorespiratory activities in a regular basis for at least six months.
* presence of negative responses on all items of the Questionnaire of Physical Activity Readiness (PAR-Q Test).

Exclusion Criteria:

* make use of medication that may interfere with the results, especially inhibitors appetites and dietary supplements.
* presence of joint problems that prevents the achievement of training.
* presence of disorders such as diabetes, dyslipidemia and anemia
* have performed intense exercise with lowers members before the training sessions.

Ages: 25 Years to 32 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura C Garay, Ph.D., Principal Investigator — University of Trás-os-Montes and Alto Douro
Locations (1):
- CEFAN, Rio de Janeiro, Rio de Janeiro, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomly assigned on August 2012 to either an interval,continuous training or control group from Sept to Dec. Tests and training were performed in a controlled laboratory condition.Tests were each separated by 24-48 h.One week before baseline they did a familiarization to submaximal test and all physiological measures.
Pre-assignment Details: Due to factors outside the present study, three individuals were removed from the program. Two individuals during maximal exercise test (VO2) showed clinical impairment test being interrupted by the doctor and the third individual presented a plantar fasciitis in the early familiarization.
Groups:
- Interval: The running training for interval group were performed on a treadmill for a period of 14 weeks, with a frequency of three times a week, lasting 20-minutes per session thus completing 46 sessions of training. The intensity and volume of training both were adapted according to the recommendations of the American College of Sports Medicine. The interval training group intensities ranged between 84-87% HRVO2peak/HRmax (vigorous intensity), 88-93%HRVO2peak/HRmax (near maximum intensity) and 94-99% HRVO2peak/HRmax (maximum intensity).
- Continuous: The running training for continuous group were performed on a treadmill for a period of 14 weeks, with a frequency of three times a week, lasting 20-minutes per session thus completing 46 sessions of training. The intensity and volume of training both were adapted according to the recommendations of the American College of Sports Medicine. The continuous group ran at an intensity of ~87%HRVO2peak/HRmax.
Period: Overall Study
Arm/Group | Interval | Continuous | Control
Started | 13 | 11 | 8
Completed | 13 | 11 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Interval: The running training for interval group were performed on a treadmill for a period of 14 weeks, with a frequency of three times a week, lasting 20-minutes per session thus completing 46 sessions of training. The intensity and volume of training both were adapted according to the recommendations of the American College of Sports Medicine. The interval training group intensities ranged between 84-87% HRVO2peak/HRmax-maximal heart rate (vigorous intensity), 88-93%HRVO2peak/HRmax (near maximum intensity) and 94-99% HRVO2peak/HRmax (maximum intensity).
- Total: Total of all reporting groups
Arm/Group | Interval | Continuous | Control | Total
Number analyzed (Participants) | 13 | 11 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (0.8) | 30.5 (1.0) | 29.1 (4.4) | 30 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 13 | 11 | 8 | 32
Region of Enrollment [Number; unit: participants]
  Brazil | 13 | 11 | 8 | 32

OUTCOME MEASURES:

1. Primary Outcome: Relative Maximal Oxygen Uptake
Description: The relative maximal oxygen uptake was taken by individual connected to a metabolic gas analyzer (VO-2000, Aerosport, Medgraphics, St. Paul, Minnesota) through which the gas samples were collected and measured each 10 seconds during the test. The participants were submitted to a ramp protocol with an initial velocity of 8.0 km/h (0% of inclination), progressive increments, a final velocity of 18 km/h (2% de inclination). The duration was equal to 10 minutes or until voluntary exhaustion.
Time Frame: Pre and post 14 weeks
Measure: Mean (Standard Deviation); unit: mL/(kg*min)
Groups:
- Continuous: The running training for continuous group were performed on a treadmill for a period of 14 weeks, with a frequency of three times a week, lasting 20-minutes per session thus completing 46 sessions of training. The intensity and volume of training both were adapted according to the recommendations of the American College of Sports Medicine.The continuous group ran at an intensity of ~87%HRVO2peak/HRmax.
Arm/Group | Interval | Continuous | Control
Number analyzed (Participants) | 13 | 11 | 8
mL/(kg*min)
  Pre VO2 | 47.8 (6.3) | 50.9 (6.0) | 49.7 (5.6)
  Post VO2 | 51.7 (5.9) | 52.8 (5.1) | 49.4 (6.4)
Statistical Analysis 1: Comparison: Interval vs Continuous vs Control; For pre-post training variables data were expressed as mean and standard deviation. Heart Rate and Blood Lactate, were by three-way ANOVA (Measure x Group x Time) with repeated measures for the factors Measure and Time. The variables absolute and relative VO2, tVO2, Body Fat, Body Mass, RPE, were made two-way ANOVAs (Group x Measure) with repeated measures on the factor Measure. Where the ANOVA was significant, the Tukey-Kramer as post-hoc was used; Test type: Superiority or Other; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: Interval vs Continuous; For pre; during (retest I 0-6weeks; retest II 0-10 weeks) and post training data were expressed as mean and standard deviation. HR and [La], were by three-way ANOVA (Measure x Group x Time) with repeated measures for the factors Measure and Time. The variables RPE, Velocity were made two-way ANOVAs (Group x Measure) with repeated measures on the factor Measure. Where the ANOVA was significant, the Tukey-Kramer as post-hoc was used. Control didn't do submaximal test for training intensities; Test type: Superiority or Other; p < 0.05, ANOVA

2. Primary Outcome: Absolute Maximal Oxygen Uptake
Description: The absolute maximal oxygen uptake was taken by individual connected to a metabolic gas analyzer (VO-2000, Aerosport, Medgraphics, St. Paul, Minnesota) through which the gas samples were collected and measured each 10 seconds during the test. The participants were submitted to a ramp protocol with an initial velocity of 8.0 km/h (0% of inclination), progressive increments, a final velocity of 18 km/h (2% de inclination). The duration was equal to 10 minutes or until voluntary exhaustion.
Time Frame: Pre and post 14 weeks
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Interval | Continuous | Control
Number analyzed (Participants) | 13 | 11 | 8
L/min
  Pre VO2 | 3.67 (0.6) | 3.89 (0.3) | 3.80 (0.5)
  Post VO2 | 4.0 (0.6) | 4.0 (0.3) | 3.7 (0.4)

3. Primary Outcome: Total Time Reaching on Maximal Test (tVO2max)
Description: The criterion for determining the total time reaching in maximal VO2 test was associated with the time immediately preceding heart rate shown a reduction of five or more beats.
Time Frame: Pre and post 14 weeks/46 sessions of training
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Interval | Continuous | Control
Number analyzed (Participants) | 13 | 11 | 8
minutes
  pre tVO2max | 9.2 (0.8) | 10.5 (1.1) | 9.6 (1.8)
  post tVO2max | 10.2 (0.7) | 10.7 (1.0) | 9.5 (1.9)

4. Primary Outcome: Heart Rate on Maximal Test
Description: The HR was collected pre and post training on maximal VO2 test. Initially, with the individual on the treadmill (Inbrasport Master Super, Porto Alegre, Brazil), electrodes (Micromed) were placed at the manubrium, right and left iliac crest for measured heart rate (HR) (derivation CM5) and were connected to an electromyography equipment (Micromed®). HR values were visualized through Elite software (Micromed Biotechnology, Brasilia, Brazil).
Time Frame: Pre and post 14 weeks at rest (5 min sitting; before start the test), during the test (to determine max), and 60s and 120s immediately after the end of the test (on sitting position)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Interval | Continuous | Control
Number analyzed (Participants) | 13 | 11 | 8
bpm
  pre HR rest | 68.8 (9.8) | 67.3 (9.6) | 65.8 (8.2)
  post HR rest | 59.3 (8.6) | 57.2 (2.1) | 64.4 (10.3)
  pre HR max | 185.3 (11.2) | 183.5 (9.4) | 190.5 (6.0)
  post HR max | 187.0 (10.6) | 185.3 (10.5) | 191.0 (8.5)
  pre HR 60s | 122.5 (19.8) | 116.3 (10) | 122.9 (22.8)
  post HR 60s | 120.9 (10.5) | 117.5 (13.3) | 123.0 (15.3)
  pre HR 120s | 110.3 (14.4) | 107.0 (9.4) | 111.6 (18.0)
  post HR 120s | 108.7 (11.1) | 108.4 (13.7) | 112.3 (13.8)

5. Secondary Outcome: Heart Rate on Submaximal Test
Description: Submaximal tests were done at the same treadmill (Treadmill® TR9100HR, Life Fitness, USA) as training.Before the test, all subjects should be able to do it at moderate-high intensity. The test began with three minutes of progressive warm-up. During the first minute, the subject maintains a light level; during the second and third minutes of the warm-up, the intensity was moderate. Starting from the fourth minute, the subject should be able to maintain a velocity for the next seven to ten minutes. This load can be adjusted as required, through verbal communication between the subject and the evaluator. The test finishes at the end of 10 minutes.The test velocity should be clearly constant at the end of the test. Heart rate were monitored and recorded at the end of each minute, e.g. 10 seconds before ending each measured minute, and the last measurement were at the end of the 10 minutes. The objective of this procedure was to identify the HR values for training intensities.
Time Frame: Pre; during (retest I 0-6weeks; retest II 0-10 weeks) and post 14 weeks/46sessions training: rest (5-min sitting; before start the test); maximal during the test (maxHRsub); 60s-120s immediately after the end of the test (on sitting position).
Population: The control group didn't do the submaximal test because it was done to determine and adjusted the training intensities during the 14 weeks.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Interval | Continuous
Number analyzed (Participants) | 13 | 11
bpm
  pre HR rest | 63.9 (6.4) | 67.2 (10.8)
  retest I HR rest | 60.8 (9.7) | 64.0 (8.5)
  retest II HR rest | 61.2 (8.8) | 59.6 (10.7)
  post HR rest | 59.8 (8.8) | 58.7 (2.6)
  pre maxHRsub | 174.8 (9.6) | 175.0 (8.3)
  retest I maxHRsub | 173.3 (10.5) | 169.8 (10.3)
  retest II maxHRsub | 174.3 (9.9) | 173.2 (10.0)
  post maxHRsub | 174.3 (7.6) | 170.1 (9.7)
  pre HR 60s | 116.2 (16.8) | 116.9 (12.5)
  retest I HR 60s | 106.5 (14.1) | 98.3 (11.6)
  retest II HR 60s | 105.5 (14.0) | 99.8 (14.4)
  post HR 60s | 103.0 (11.3) | 100.7 (12.7)
  pre HR 120s | 98.9 (14.8) | 102.3 (9.2)
  retest I HR 120s | 90.5 (13.4) | 87.5 (10.5)
  retest II HR 120s | 91.9 (17.4) | 90.8 (12.3)
  post HR 120s | 93.8 (11.9) | 89.9 (9.3)

6. Secondary Outcome: Blood Lactate on Submaximal Test
Description: Capillary blood samples (25 µl) were obtained from the finger of each subject during all tests and the [La] were measured using an (Accutrend®Plus Roche Diagnostics Gesellschaft mit beschränkter Haftung , Mannheim, Germany). The measuring range was 0.8-22 mM. The sample is collecting (Accu-Chek® Softclix) and first applied to a coded yellow test strip (Accutrend Blood Measure-Roche) with a reagent chemical substance. Blood was added to the strip by letting it drip from a finger; in accordance with the instrument's instructions we never let the finger touch the strip's pad in order to exclude any possible interference due to the sweat.
Time Frame: Pre; during (retest I 0-6weeks; retest II 0-10 weeks) and post 14 weeks/46 sessions training: rest (5-min sitting; before start the test); 1-3-5 minutes immediately after the end of the test (on sitting position).
Population: The control group didn't do the submaximal test because it was done to determine and adjusted the HR training intensities and also collected [La] on rest and after submaximal effort during 14 weeks of training.
Measure: Mean (Standard Deviation); unit: mmol*L^-1
Arm/Group | Interval | Continuous
Number analyzed (Participants) | 13 | 11
mmol*L^-1
  pre [La] rest | 2.59 (0.33) | 2.40 (0.22)
  retest I [La] rest | 2.66 (0.57) | 2.45 (0.39)
  retest II [La] rest | 2.42 (0.40) | 2.25 (0.44)
  post [La] rest | 2.81 (0.39) | 2.56 (0.50)
  pre [La] 1-min | 7.41 (2.28) | 9.39 (2.30)
  retest I [La] 1-min | 7.52 (1.81) | 6.94 (1.75)
  retest II [La] 1-min | 8.14 (2.34) | 7.89 (1.50)
  post [La] 1-min | 8.12 (2.37) | 7.69 (2.10)
  pre [La] 3-min | 6.96 (2.43) | 8.80 (2.48)
  retest I [La] 3-min | 6.52 (1.93) | 5.65 (1.05)
  retest II [La] 3-min | 7.50 (2.23) | 7.00 (1.39)
  post [La] 3-min | 7.52 (2.25) | 7.07 (2.02)
  pre [La] 5-min | 5.85 (2.33) | 7.21 (3.18)
  retest I [La] 5-min | 5.80 (1.74) | 5.22 (1.35)
  retest II [La] 5-min | 6.91 (2.34) | 6.49 (1.27)
  post [La] 5-min | 6.79 (2.03) | 6.49 (2.03)

7. Secondary Outcome: Submaximal Velocity [Vsub]
Description: Submaximal tests were done at the same treadmill (Treadmill® TR9100HR, Life Fitness, USA) as training.Before the test, all subjects should be able to do it at moderate-high intensity. The test began with three minutes of progressive warm-up. During the first minute, the subject maintains a light level; during the second and third minutes of the warm-up, the intensity was moderate. Starting from the fourth minute, the subject should be able to maintain a velocity for the next seven to ten minutes. This load can be adjusted as required, through verbal communication between the subject and the evaluator. The test finishes at the end of 10 minutes. The test velocity should be clearly constant at the end of the test. Values of velocity were monitored and recorded at the end of each minute, e.g. 10 seconds before ending each measured minute, and the last measurement were at the end of the 10 minutes. The objective of this procedure was to identify the value of that speed has stabilized.
Time Frame: Pre; during (retest I 0-6weeks; retest II 0-10 weeks) and post 14 weeks/46sessions of training
Population: The control group didn't do the submaximal test because it was done to determine and adjusted the HR training intensities and also collected [Vsub] during submaximal effort.
Measure: Mean (Standard Deviation); unit: km/h
Arm/Group | Interval | Continuous
Number analyzed (Participants) | 13 | 11
km/h
  pre [Vsub] | 13.2 (2.0) | 13.9 (1.4)
  retest I [Vsub] | 13.4 (0.8) | 13.7 (1.6)
  retest II [Vsub] | 13.9 (0.6) | 14.4 (1.1)
  post [Vsub] | 13.9 (0.8) | 13.9 (0.9)

8. Secondary Outcome: Rate of Perceived Exertion (RPE) on Submaximal Test
Description: The RPE was collected at submaximal test (see description of test on outcome measure "HR at submaximal test"). Relative to overall feelings were collected by Category Ratio Scale (CR10) during the last 15 s of each stage using the Borg category (0 - 10) scale. Instructions for RPE were that "0" corresponds to rest, and "9 - 10" corresponds to maximal exertion. This verbal procedure was explained before initiating exercise.
Time Frame: Pre; during (retest I 0-6weeks; retest II 0-10 weeks) and post 14 weeks/46sessions training
Population: The control group didn't do the submaximal test because it was done only for determine and adjusted the training intensities.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interval | Continuous
Number analyzed (Participants) | 13 | 11
units on a scale
  pre RPE | 6 (1) | 6 (2)
  retest I RPE | 6 (1) | 5 (1)
  retest II RPE | 6 (2) | 6 (2)
  post RPE | 7 (2) | 7 (1)

9. Primary Outcome: Blood Lactate Concentrations on Maximal Test
Description: Capillary blood samples (25 µl) were obtained from the finger of each subject during all tests and the [La] were measured using an (Accutrend®Plus Roche Diagnostics Gesellschaft mit beschränkter Haftung , Mannheim, Germany). The measuring range was 0.8-22 millimole (mM). The sample is collecting (Accu-Chek® Softclix) and first applied to a coded yellow test strip (Accutrend Blood measure-Roche) with a reagent chemical substance. Blood was added to the strip by letting it drip from a finger; in accordance with the instrument's instructions. The finger never touched the strip's pad in order to exclude any possible interference due to the sweat. All [La] were collected by a single, experienced investigator.
Time Frame: Pre and post 14 weeks/46sessions on rest (5 min sitting position; before start the test); 1-3-5 min immediately after the end of the test (on sitting position).
Measure: Mean (Standard Deviation); unit: mmol*L^-1
Arm/Group | Interval | Continuous | Control
Number analyzed (Participants) | 13 | 11 | 8
mmol*L^-1
  pre [La] rest | 2.55 (0.38) | 2.40 (0.20) | 2.36 (0.23)
  post [La] rest | 2.73 (0.39) | 2.29 (0.45) | 2.68 (0.23)
  pre [La] 1-min | 12.03 (2.89) | 12.21 (2.49) | 13.41 (1.54)
  post [La] 1-min | 13.14 (2.57) | 13.23 (1.57) | 13.30 (1.39)
  pre [La] 3-min | 11.42 (2.23) | 11.97 (2.90) | 12.88 (1.56)
  post [La] 3-min | 12.66 (2.50) | 12.88 (1.65) | 13.44 (1.56)
  pre [La] 5-min | 9.74 (3.40) | 11.5 (2.74) | 12.26 (1.74)
  post [La] 5-min | 13 (2.58) | 12.9 (1.49) | 13.45 (1.40)

10. Primary Outcome: Body Mass (BM)
Description: To measure body mass Filizola scales with a stadiometer was used.
Time Frame: Body Mass was collected pre and post training
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Interval | Continuous | Control
Number analyzed (Participants) | 13 | 11 | 8
kg
  pre BM | 77.6 (13.5) | 76.6 (3.7) | 76.4 (10.9)
  post BM | 77.5 (13.7) | 76.1 (4.4) | 76.0 (11.1)

11. Primary Outcome: Rate of Perceived Exertion (RPE) on Maximal Test
Description: The RPE was collected at maximal test (see description of test on outcome measure "Maximal Oxygen Uptake"). Relative to overall feelings were collected by Category Ratio Scale (CR10) during the last 15 s of each stage using the Borg category (0 - 10) scale. Instructions for RPE were that "0" corresponds to rest, and "9 - 10" corresponds to maximal exertion. This verbal procedure was explained before initiating exercise.
Time Frame: Pre and post 14 weeks/46 sessions of training
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interval | Continuous | Control
Number analyzed (Participants) | 13 | 11 | 8
units on a scale
  pre RPE | 8.9 (0.9) | 9.5 (0.9) | 9.2 (1.0)
  post RPE | 8.8 (1.5) | 9.0 (1.3) | 9.0 (0.9)

12. Primary Outcome: Fat Mass (%)
Description: The subjects underwent a set of anthropometric assessments, which followed the norms of the International Society for Advancement of Kinanthropometry. The fat mass was calculated by percentage using the equation proposed by Jackson and Pollock (1978) from seven skinfold measurement. To measure the skinfolds, a Sanny Professional Skinfold Caliper was used.
Time Frame: Pre and post 14 weeks/46 sessions of training
Measure: Mean (Standard Deviation); unit: Fat Mass %
Arm/Group | Interval | Continuous | Control
Number analyzed (Participants) | 13 | 11 | 8
Fat Mass %
  pre | 14.3 (6.0) | 11.9 (3.9) | 12.5 (4.9)
  post | 14.9 (5.6) | 13.6 (5.1) | 13.4 (4.7)

ADVERSE EVENTS:
Arm/Group | Interval | Continuous | Control
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 0/8
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No